CLINICAL TRIAL: NCT05150301
Title: Study of the Short-term Mortality and Morbidity of Newborns Born at a Gestational Age <32 Weeks of Amenorrhea Outside a Level III Maternity Hospital in Alsace
Brief Title: Study of the Short-term Mortality and Morbidity of Newborns Born at a Gestational Age <32 Weeks of Amenorrhea
Acronym: OutBorn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8425
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Premature Birth
Keywords: Premature Birth; Outborn; Newborns; Gestational age
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An "outborn" birth is a premature birth that occurs in an unsuitable level center at the end of the child (unlike "inborn" births).

This study aims to describe the morbidity and mortality of very premature newborns (gestational age less than 32 weeks of amenorrhea) born outside a maternity hospital of appropriate level between January 1, 2016 and December 31, 2020, and assessment of the preventable or non-preventable nature of these so-called "outborn" births.

The aim of this research is to write down the short-term mortality and morbidity of newborns born at a gestational age <32 weeks of amenorrhea outside a level III maternity hospital in Alsace between January 1, 2016 and December 31, 2020.

ELIGIBILITY:
Inclusion criteria:

- Newborn under 32 weeks of amenorrhea at the time of birth, born in Alsace in one of the level I, IIa, or IIb maternity hospitals, between January 1, 2016 and December 31, 2020

Exclusion criteria:

- Fetal death in utero

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn under 32 weeks of amenorrhea at the time of birth, born in Alsace in one of the level I, IIa, or IIb maternity hospitals, between January 1, 2016 and December 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Study of the short-term mortality and morbidity of newborns born at a gestational age <32 weeks of amenorrhea | Files analysed retrospectively from January 01, 2016 to December 31, 2010 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Benoit ESCANDE, MD, Principal Investigator — Service de Réanimation Néonatale - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Réanimation Néonatale - Hôpitaux Universitaires de Strasbourg, Strasbourg, France